CLINICAL TRIAL: NCT06061614
Title: A Clinical Study for the Safety and Efficacy of IV Infusion of NGGT002 in the Treatment of Phenylketonuria
Brief Title: Safety and Efficacy Study of NGGT002 in PKU Adult Subjects
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NGGT002-P-2202
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Phenylketonurias
Keywords: PAH Deficiency
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Intervention Model Description: single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose level 1 (Experimental): Dose level 1 will be administered
  Interventions: Genetic: NGGT002
- Dose level 2 (Experimental): Dose level 2 will be administered
  Interventions: Genetic: NGGT002
- Dose level 3 (Experimental): Dose level 3 will be administered
  Interventions: Genetic: NGGT002

INTERVENTIONS:
Genetic: NGGT002 — NGGT002

SUMMARY:
This investigator initiated trial is an open-label, dose escalation study to evaluate the safety, tolerability and efficacy of NGGT002, an AAV derived investigational gene therapy product expressing human PAH enzyme in adult Phenylketonuria (PKU) subjects with PAH deficiency. All participants will receive a single administration of NGGT002 and will be followed for safety and efficacy for 5 years.

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of NGGT002 gene therapy with three dose cohorts in adult subjects with diagnosis of PKU characterized by PAH deficiency with confirmed PAH gene mutations. NGGT002 will be administered through intravenous infusion. Dose escalation will be initiated from the low dose of NGGT002. After evaluating the safety and efficacy data, a decision will be made regarding the cohort expansion or the escalation to the next dose level. The same process will be followed for subsequent dose cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign informed consent form;
* Male and female subjects with diagnosis of PKU caused by confirmed PAH mutation as per the "Clinical Practice Guidelines for Phenylketonuria 2020";
* Age ≥ 18 years;
* Phe concentration ≥ 600 μmol/L at screening and ≥ 600 μmol/L at least once within 2 years prior to screening;
* Subjects who are willing and able to maintain their baseline diet throughout the study, regardless of phenylalanine restriction, except at the investigator's request;

Exclusion Criteria:

* Presence of anti-AAV8 neutralizing antibody
* Prior gene therapy
* Positive hepatitis B virus surface antigen, hepatitis C virus antibody, anti-human immunodeficiency virus antibody or treponema pallidum-specific antibody
* Hepatic function abnormal: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 × ULN; alkaline phosphatase (ALP) > 1.5 × ULN; total bilirubin (TBil) > 1.5 × ULN; international normalized ratio (INR) > 1.3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | Week 52
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) from baseline to week 52 (W52)

SECONDARY OUTCOMES:
plasma Phe levels | W12, W28, W52
  Change from baseline in mean plasma Phe levels

OTHER OUTCOMES:
total protein intake | W12, W28, W52
  Change from baseline in total protein intake

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No